CLINICAL TRIAL: NCT02656524
Title: Effectiveness of Stivarga (Regorafenib) for Patients With Metastatic Colorectal Cancer in the Hungarian Real World Setting
Brief Title: Stivarga Real Life Evidence in Hungary
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18686
Record Dates: First submitted 2015-12-21; First posted 2016-01-15 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Colorectal Neoplasms
Keywords: Metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort1/Regorafenib: All patients with at least 1 treatment with regorafenib
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — Product is used in accordance with SmPC

SUMMARY:
The study aims to evaluate use of regorafenib in clinical practice in Hungary. The study should provide information about clinical characteristics of Hungarian regorafenib patients as well as information about safety and efficacy of regorafenib in Hungarian patients with metastatic colorectal cancer. This much needed data is required by the National Health Insurance Fund in order to accept regorafenib into the regular reimbursement system. This study is proposed to be based on patient data from the Hungarian National Health Insurance Fund's Database. Data to be analyzed includes patient demography and baseline tumor characteristics, overall survival, time to treatment failure, duration of treatment, average dose and dose modifications, and adverse events. Further, treatment costs will be estimated.

ELIGIBILITY:
Inclusion Criteria:

* Using the National Health Insurance Database, patients will be included in this retrospective data analysis if they had at least one dose of regorafenib treatment cycle (=28 days).

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be all patients who met the criteria within the SmPC. Using the National Health Insurance Database, patients will be included in this retrospective data analysis if they had at least one dose of regorafenib treatment cycle.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Length of treatment for each treatment episode | Retrospective analysis of 2 year period
  The length of each treatment episode will be calculated based on the duration between the initiation date of a treatment episode and the end date of the same treatment episode
Progression Free Survival (PFS) | Retrospective analysis of 2 year period
  PFS will be defined as days between start of the therapy and the date of the medical doctors opinion about progression (confirmed by radiology or clinical assessment)
Overall Survival (OS) | Retrospective analysis of 2 year period
Number of participants with treatment emergent adverse events as a measure of safety and tolerability | Retrospective analysis of 2 year period

SECONDARY OUTCOMES:
Resource utilization per patient | Retrospective analysis of 2 year period
  Costs per patient for the reimbursed healthcare service e.g. inpatient care, outpatient visit, emergency departement visit, pharmaceutical dispensing

OTHER OUTCOMES:
Time to treatment failure (TTF) | Retrospective analysis of 2 year period
  Time to treatment failure is defined as days between the first drug delivery to the health care provider and date of treatment discontinuation due to any reason, including death
Time to progression (TTP) | Retrospective analysis of 2 year period
  Time to progression is defined as days between the first drug delivery to the health care provider and the date of progression defined by the medical doctor
Characteristics of patients with better response | Retropsective analysis of 2 year period
  Patients with "better response" are defined as receiving more cycles of regorafenib treatment than the median number of cycles (2 cycles). Their distribution is analyzed by KRAS status, by the location of the primary tumour, by age, by prior cancer therapies and by location of metastases.
Time frame between the baseline computed tomography and the first drug delivery | Retrospective analysis of 2 year period
  Time frame between the date of the baseline computed tomography (CT) and the date of the first drug delivery to the health care provider

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Budapest, Hungary